CLINICAL TRIAL: NCT03290235
Title: The Extension Study of Phase IV Clinical Trial of Pegylated Somatropin (PEG Somatropin) to Treat Growth Retardation Caused by Endogenous Growth Hormone Deficiency in Children
Brief Title: Extension Study of Pegylated Somatropin to Treat Growth Retardation Caused by Endogenous Growth Hormone Deficiency in Children
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Changchun GeneScience Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GenSci 045 CT-Extension Period
Record Dates: First submitted 2017-09-19; First posted 2017-09-21 (Actual); Last update posted 2017-12-12 (Actual); Status verified 2017-09

CONDITIONS: Growth Retardation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PEG-somatropin-1 (Experimental): Dosage 0.2mg/kg/w
  Interventions: Drug: PEG-somatropin
- PEG-somatropin-2 (Experimental): Dosage 0.1-0.2mg/kg/w
  Interventions: Drug: PEG-somatropin

INTERVENTIONS:
Drug: PEG-somatropin — Pegylated somatropin, injection, 54IU/9.0mg/1.0ml/kit
  Other Names: Jintrolong®

SUMMARY:
1. To further evaluate the safety and efficacy of PEG-Somatropin in the treatment of children with growth hormone deficiency for a relatively long period
2. To explore the factors influencing the efficacy of PEG-Somatropin and to establish the height prediction model based on Chinese children with short stature, and to provide the basis and guidance for standard and reasonable long-term clinical application of PEG-Somatropin.

ELIGIBILITY:
Inclusion Criteria:

* Children has completed all visits and therapy in previous phase IV study;
* Investigators evaluate subjects could continue growth hormone therapy;
* Subjects is willing and able to cooperate to complete scheduled visits, treatment plans and laboratory tests and other procedures, to sign informed consent.

Exclusion Criteria:

* Children with epiphyseal closure;
* Children is near the adule final height, that is, growth rate≤ 2 cm / year or bone age ≥ 14 years old for girls, bone age ≥ 16 years old for boys;
* Dysfunction of liver and kidney (ALT> 2 times the upper limit of normal, Cr> upper limit of normal);
* Patients with known hypersensitivity to PEG-Somatropin or Somatropin or any other components of the study product;
* Patients with severe cardiopulmonary or hematological diseases, a current or past history of malignant tumors, immunodeficiency diseases, or mental diseases;
* Patients with diabetics;
* Patients with congenital bone dysplasia or scoliosis;
* Patients took drugs that would influence the efficacy and safety of PEG-Somatropin after phase IV study and before screening for this extension study;
* Other conditions in which the investigator preclude enrollment into the study.

Ages: 42 Months to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 1500 (Estimated)
Dates: Start 2017-03-01 (Actual); Primary Completion 2020-10 (Estimated); Study Completion 2021-09 (Estimated)

PRIMARY OUTCOMES:
Ht SDSca (Height standard deviation score for chronological age) | Baseline, every 13 weeks until 130 weeks
  Calculated by dividing the difference between the actual height of a patient and the mean height of the population for that chronological age by the standard deviation (SD) of the height of the population for that chronological age

SECONDARY OUTCOMES:
Ht SDSBA (Height standard deviation score for bone age) | Baseline, every 13 weeks until 130 weeks
Yearly growth velocity | Baseline, every 13 weeks until 130 weeks
IGF-1 SDS (Standard deviation score of insulin-like growth factor-1) | Baseline, every 13 weeks until 130 weeks
Bone age | Baseline, 26 weeks, 52 weeks, 78 weeks, 104 weeks, 130 weeks
Near final height for some subjects | Baseline, every 13 weeks until 130 weeks
  When yearly growth velocity of some subject is no more than 2cm/year.

CONTACTS AND LOCATIONS:
Locations (1):
- TongJi hospital affiliated to TongJi medical college of HuaZhong university of Science & Teconology, Wuhan, Hubei, China

REFERENCES:
- [Derived] Hou L, Huang K, Gong C, Luo F, Wei H, Liang L, Du H, Zhang J, Zhong Y, Chen R, Chen X, Pan J, Jin X, Zeng T, Liao W, Liu D, Lan D, Zhu S, Dong Z, Ma H, Yang Y, Xiong F, Lu P, Cheng S, Gu X, Jin R, Liu Y, Wu J, Xu X, Chen L, Dong Q, Pan H, Su Z, Liu L, Luo X, Ni S, Chen Z, Hu Y, Wang C, Liu J, Liu L, Lu B, Wang X, Wang Y, Yang F, Zhang M, Cao L, Liu G, Yao H, Zhan Y, Dai M, Li G, Li L, Liu Y, Wang K, Xiao Y, Zhang X, Dong J, Gu Z, Ying L, Huang F, Liu Y, Liu Z, Ye J, Zhao D, Hu X, Jiang Z, Ye K, Zhu H, Chen S, Chen X, Wan N, Xu Z, Yin Q, Zhang H, Huang X, Yin J, Zhang H, Li P, Yin P, Fu J, Luo X. Long-term Pegylated GH for Children With GH Deficiency: A Large, Prospective, Real-world Study. J Clin Endocrinol Metab. 2023 Jul 14;108(8):2078-2086. doi: 10.1210/clinem/dgad039. PMID 36669772